CLINICAL TRIAL: NCT02322385
Title: Mutational Types and Phenotypes Relationship in Autosomal Dominant Polycystic Kidney Disease
Brief Title: Clinical Implications of DNA Analysis on ADPKD
Acronym: DNAAA
Status: Completed | Type: Observational
Sponsor: Kyorin University (Other)
Collaborators: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Eiji Higashihara, MD, Professor of Department of Polycystic Kidney Research, Kyorin University School of Medicine., Kyorin University
Other Study IDs: Kyorin-PKD-1
Record Dates: First submitted 2014-01-24; First posted 2014-12-23 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Autosomal Dominant Polycystic Kidney Disease
Keywords: Autosomal Dominant Polycystic Kidney Disease; PKD 1 gene; PKD 2 gene; Truncational mutation; Hypomorphic mutation
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No

SUMMARY:
Autosomal dominant polycystic kidney disease (ADPKD) is an inherited disease. We plan DNA analysis using the next generation sequencer (NGS) and examine the relationship between mutational types and clinical phenotypes. The accuracy of DNA analysis with NGS is tested by Sanger's method. The kidney and life survival curves will be compared between PKD1, PKD2 and non-ADPKD family members.

DETAILED DESCRIPTION:
80 unrelated patients with ADPKD attending to the Kyorin University Hospital whose clinical data are compiled. DNA analysis is performed at Otsuka Pharmaceutical Laboratory.

Clinical data include total kidney volume (TKV), TKV slope, eGFR, eGFR slope and other clinically relevant data.

ELIGIBILITY:
Inclusion Criteria:

* The unrelated patients with ADPKD.

Exclusion Criteria:

* The patients whose clinical data are not compiled.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients with ADPKD visiting Kyorin university hospital over two years. The patients whose clinical data including total kidney volume (TKV), eGFR, QOL data and other relevant clinical data are available will be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2014-01; Primary Completion 2016-12-31 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
The relationship between mutational types and phenotypes | Depends on the observational period at least more than one year.
  * Total Kidney Volume (TKV) measured by MRI and its slope.
  * Total Liver Volume (TLV) measured by MRI and its slope.
  * GFR estimated by plasma creatinine and cystatin C (eGFR).
  * Other clinical data, such as QOL scores and ADPKD-related symptoms.

SECONDARY OUTCOMES:
Identify the efficacy of next generation sequencing method | One year.
  * Compatibility of sequence results between two NGSs.
  * Compatibility of sequence results between NGS and Sanger's method.

OTHER OUTCOMES:
The relationship between mutational types and phenotypes; | One year.
  • The radiologic findings of intracranial aneurysm and cerebral arteries.

CONTACTS AND LOCATIONS:
Overall Officials: Eiji Higashihara, MD, Study Chair — Department of Polycystic Kidney Research, Kyorin University School of Medicine
Locations (2):
- Japan (2):
  - Department of Polycystic Kidney Research, Kyorin University School of Medicine, Mitaka, Tokyo
  - Department of Urology, Kyorin University Hospital, Mitaka, Tokyo

REFERENCES:
- [Derived] Higashihara E, Horie S, Kinoshita M, Harris PC, Okegawa T, Tanbo M, Hara H, Yamaguchi T, Shigemori K, Kawano H, Miyazaki I, Kaname S, Nutahara K. A potentially crucial role of the PKD1 C-terminal tail in renal prognosis. Clin Exp Nephrol. 2018 Apr;22(2):395-404. doi: 10.1007/s10157-017-1477-7. Epub 2017 Oct 5. PMID 28983800